CLINICAL TRIAL: NCT07154277
Title: Abdominal Midline Incisional Closure With Small Bites Vs Large Bites in Emergency Settings
Brief Title: Small Bites Vs Large Bites Abdominal Midline Incisional Closure
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2888
Record Dates: First submitted 2024-07-12; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-12

CONDITIONS: Suture Techniques; Wound Closure Techniques; Laparotomy/Standerds; Surgical Wound Dehiscence; Incisional Hernia/Prevention and Control; Surgical Wound Infection
Keywords: midline abdominal closure; emergency laparotomy; small bite closure; large bite closure; wound closure
MeSH Terms: conditions — Surgical Wound Dehiscence; Incisional Hernia; Surgical Wound Infection

STUDY DESIGN:
Intervention Model Description: Patients are randomly categorized into two different groups and treated differently and outcomes are assessed in the same manner in both groups.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Masking is done only for outcome assessor as it is not possible for others to be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Large Bite Closure of midline laparotomy wound (Active Comparator): Standard closure: Suture bite should be 1 cm away from wound margin and 1 cm apart from the previous suture bite
  Interventions: Procedure: Large bite closure
- Small Bite Closure of midline laparotomy wound (Experimental): Small Bite closure: Suture bite should be 0.5 cm away from wound margin and 0.5 cm apart from the previous suture bite
  Interventions: Procedure: Small bite closure

INTERVENTIONS:
Procedure: Small bite closure — Small bite suturing is small tissue bite of 0.5cm depth x 0.5cm travel x 0.5cm apart, on the aponeurosis away from midline using Prolene 2/0
  Other Names: small bite suturing technique; small bite suture; 0.5*0.5*0.5 suturing technique
  Arms: Small Bite Closure of midline laparotomy wound
Procedure: Large bite closure — Large bite closure is defined as tissue bite of 1cm depth x 1 cm travel x 1cm apart, on the aponeurosis away from midline using Prolene 0
  Other Names: Large bite suturing technique; Large bite suture; Large suturing technique
  Arms: Large Bite Closure of midline laparotomy wound

SUMMARY:
The goal of this trial is to compare the effectiveness of small bite versus large bite abdominal incision closure in emergency settings. It will also evaluate the safety and outcomes of each technique. The main questions it aims to answer are:

Does small bite closure reduce the incidence of superficial surgical site infections (SSI), wound dehiscence, and incisional hernia compared to large bite closure? What are the associated complications of each closure technique?

Participants will:

Undergo either a small bite or large bite abdominal incision closure during emergency laparotomy Visit the clinic for follow-up assessments at 7 days, 15 days, 1 month, 3 months, and 6 months post-operatively Have their wound healing and complications documented and analyzed during respective visits.

DETAILED DESCRIPTION:
Background Wound site complications continue to be a major detrimental factor in surgical healthcare around the globe and are a major concern for general surgeons due to the associated morbidity and mortality. Superficial Surgical Site Infection (SSI) is defined as an infection related to a surgical procedure that occurs near the surgical site within 30 days following surgery (or up to 90 days following surgery where an implant is involved). The incidence of such complications is generally higher in emergency laparotomies compared to elective cases. Surgical technique plays a key role in the integrity of the post-operative wound, and among the numerous factors that influence wound healing, it is the only one under the direct control of the surgeon. The midline incision is the most commonly used surgical incision for emergency laparotomy as it provides quick, wide exposure and avoids damage to nerves, muscles, and the blood supply of the abdominal wall. Closure of the midline wound has traditionally been performed using a mass fashion or large bite technique with a running suture, but recently a new technique of small bite closure has been proposed.

Hypothesis The hypothesis is that small bite closure will have better outcomes than large bite closure in terms of reducing acute wound failure.

Objective This study aims to compare the effectiveness of small bite abdominal incision closure with large bite closure in patients undergoing emergency laparotomy at a tertiary hospital in Karachi, Pakistan.

Materials and Methods

A single-blinded randomized comparative trial will be conducted at Civil Hospital, a tertiary hospital in Karachi, Pakistan. A total of 200 participants will be recruited for this study, with equal participants divided into two groups. Patients undergoing emergency laparotomies will be randomly assigned to one of two groups:

Group A: Participants will undergo large bite closure. Group B: Participants will undergo small bite closure. Participants will be followed up at 7 days, 15 days, 1 month, 3 months, and 6 months postoperatively to assess for complications. Data collection will be done using a single-blinded, block randomization method, where each participant will be assigned a unique code.

Operational Definitions Effectiveness: Defined by the incidence of superficial SSI, wound dehiscence, and incisional hernia in the two study groups.

Superficial SSI: An infection near the surgical site within 30 days of surgery (or up to 90 days with an implant) involving only skin or subcutaneous tissue. Diagnosed by purulent drainage, isolated organisms from an aseptically obtained culture, or symptoms like pain, tenderness, localized swelling, redness, heat, and diagnosis by a surgeon or attending physician.

Wound Dehiscence: Partial or total separation of previously approximated wound edges due to failed wound healing.

Incisional Hernia: An abnormal protrusion of abdominal contents through the weakness in the abdominal wall at the incision site.

Large Bite Closure: Tissue bite of 1cm depth, 1cm travel, and 1cm apart, using Prolene 0.

Small Bite Closure: Tissue bite of 0.5cm depth, 0.5cm travel, and 0.5cm apart, using Prolene 2/0.

Jenkin's Rule: A 4:1 suture to wound ratio. Data Collection and Analysis Data will be collected through a structured Performa and analyzed using the latest version of SPSS. The analysis will focus on comparing the incidence of superficial SSI, wound dehiscence, and incisional hernia between the two groups, providing insights into the effectiveness of each closure technique.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages in between 18-60 year old
* All emergency laparotomies (Except trauma)

Exclusion Criteria:

* Previous surgery with midline incision
* Pregnancy
* Current immunosuppressive or chemotherapy
* Previous incisional hernia after midline incision

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Wound Dehiscence | 1 month
  Wound dehiscence as seen by the surgeon.
Number of participants with Surgical Site Infections | 1 month
  As per CDC guidelines and seen by the surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Omer Bin Khalid Jamil, Principal Investigator — Ruth K.M. Pfau Civil Hospital Karachi
Locations (1):
- Dr. Ruth K. M. Pfau Civil Hospital Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No